CLINICAL TRIAL: NCT03551795
Title: Clinical Research on Comprehensive Treatment of Tuberculosis With Malignant Solid Tumor
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xiaoyan Zhang (Other Government)
Responsible Party: Sponsor-Investigator, Xiaoyan Zhang, Principal Investigator, Shanghai Public Health Clinical Center
Organization: Shanghai Public Health Clinical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iNKT20180427V1.1
Record Dates: First submitted 2018-05-01; First posted 2018-06-11 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Malignant Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): The eligible patient receive the experimental infusion of iNKT cells.
  Interventions: Biological: Infusion of iNKT cells

INTERVENTIONS:
Biological: Infusion of iNKT cells — The eligible patients receive twice infusions of iNKT cells(1E8~1E10) in one course of treatment.

SUMMARY:
Invariant Natural killer T (iNKT) cells are a unique subset of lymphocytes that express homogeneous TCR recognizing KRN7000 which was up-regulated by many kinds of cancer cells.The hypothesis of the investigators is that immunotherapy strategy of infusion of iNKT cells may resist inflection and decrease the tumor burden and improve overall survival. The purpose of this study is to assess the safety and efficacy of treatment of tuberculosis with malignant solid tumor by infusing of iNKT cells.

DETAILED DESCRIPTION:
Treatment of tuberculosis with malignant solid tumor is great unsolved challenge to the physicians. Efficacy of conventional treatment, such as surgery, radiotherapy and chemotherapy is limited. AS novel therapy, immunotherapy shows great prospects.

Human iNKT cells can directly lysis tumor cells by a perforin-dependent mechanism,and intracellular granzyme B expression may also potentiate cell killing. Tumor cells expressing CD1d may be especially susceptible to direct NKT cell lysis. iNKT cells play important role in immune regulation by secreting various cytokines. Expansion method of iNKT cells in vitro is developed as published in the patent of the investigators. Infusion of iNKT cells has been proved safe in mice.

In this clinical trial, the safety and efficacy of the immunotherapy of infusion of iNKT cells are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytologically diagnosis of tuberculosis with malignant solid tumor
* Patients' tumor tissue (formalin-fixed, paraffin-embedded) must be sufficient for diagnosis of cancer by a certified Laboratory of Pathology
* Laboratory values within the following ranges prior to receiving treatment of study agent: Hemoglobin≧8.0 g/dL, Neutrophils count≧1E9/L, Lymphocytes count≧lower limit of institutional normal, Platelet count≧50E9/L, Serum creatinine≦2.0 mg/dL, Serum bilirubin≦2 x upper limit of institutional normal, AST/ALT≦2 x upper limit of institutional normal
* No dyspnea at rest. Oxygen saturation ≥90% on room air
* No genetic disease
* Fertile females/males must consent to use contraceptives during participation of the trial. Women of child bearing potential must have a negative pregnancy test prior to receiving treatment of study agent within 7 days
* Patients must have a Karnofsky performance status greater than or equal to 80%
* Able and willing to give witnessed, written informed consent form prior to receiving any study related procedure
* Agrees to participate in long-term follow-up for up to 1 years, if received NKT infusion

Exclusion Criteria:

* Organ dysfunction,such as significant cardiovascular disease, myocardial infarction within the past six months, unstable angina, coronary angioplasty within the past six months, uncontrolled atrial or ventricular cardiac arrhythmias; Child-Pugh C; Renal function failure or uremia; Respiratory failure; Disturbance of consciousness; Renal failure.
* Suffering from lymphoma or leukemia
* Serious infections requiring antibiotics, bleeding disorders
* Patients with myelodysplastic syndrome (MDS)
* History of immunodeficiency disease or autoimmune disease
* Positive HIV antigen and antibody, Hepatitis B surface antigen and Hepatitis C PCR within 21 days prior to enrollment
* Within concurrent chemotherapy
* Concurrent other medical condition that would prevent the patient from undergoing protocol-based therapy
* Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dose of study agent
* Pregnant or breast-feeding patients
* Can't give informed consent
* Lack of availability for follow-up assessment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 4 months post-infection
  Change of target focus confirmed by CT or MRI

SECONDARY OUTCOMES:
Incidence of adverse events related to the infusion of cells | 28 days post-infusion
  The incidence of adverse events following infusion of iNKT cells

OTHER OUTCOMES:
Progression-Free Survival (PFS) | Approximately 1 years after the treatment
  Progression-Free Survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Qing J Xu, Ph.D, Study Chair — Shanghai Public Health Clinical Center, Fudan University, 2901 Caolang Road, Jin Shan, Shanghai 201508, P.R. China
Locations (1):
- Shanghai Public Health Clinical Center, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No